CLINICAL TRIAL: NCT02050984
Title: A Prospective Study on the Effects of Bariatric Surgery on Blood Pressure in Patients With Obesity and Diabetes
Brief Title: Effect of Bariatric Surgery on Blood Pressure
Acronym: BASBP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhiming Zhu (Other)
Responsible Party: Sponsor-Investigator, Zhiming Zhu, Director of the Dept. of Hypertension & Endocrinology, Third Military Medical University
Organization: Third Military Medical University (Other)
Other Study IDs: BASBP; 2012CB517805 (Other Grant/Funding Number: National Basic Research Program of China)
Record Dates: First submitted 2014-01-25; First posted 2014-01-31 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Obesity; Diabetes
Keywords: Obesity; Hypertension; Bariatric Surgery; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Bariatric surgery is generally recommended for obese people with a body mass index (BMI) of at least 40kg/m2, and for people with BMI 35 kg/m2 and serious coexisting medical conditions such as diabetes. A variety of studies showed that it cause significant weight loss, recovery from diabetes and improvement in cardiovascular risk factors, such as blood pressure. The recent guidelines suggest that patients with a BMI of more than 30 kg/m2 with co morbidities is a candidate for bariatric surgery. However, the patients with diabetes in Chinese has lower BMI than that in west country. Therefore, this research is designed to observe whether bariatric surgery reduce blood pressure in patients with diabetes and relatively lower BMI.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 60 years old.
* Type 2 Diabetes diagnosis defined according to WHO 2006 guideline.
* Body mass index between 25.0 and 39.9 kg/m2.

Exclusion Criteria:

* Hypertension ≥ 180/120 mmHg;
* Type 1 diabetes, other types of diabetes or gestational diabetes;
* Acute complications of diabetes;
* Cerebrovascular diseases in the last 6 months.
* Cardiovascular diseases (myocardial infarction, angina, cardiac failure) in the last 6 months.
* Baseline psychiatric disorders: schizophrenia, bipolar disorder, severe depression, psychosis.
* Renal diseases: diabetic nephropathy, creatinine clearance < 30 ml/min.
* Advanced peripheral arterial disease
* Atrophic gastritis
* Alcoholism or use of illicit drugs
* Previous laparotomy
* Severe hepatic disorders
* Pregnancy or women not using effective contraceptive methods.
* Recent neoplasm (< 5 years)
* Immunosuppressant drugs
* Unable to understanding and follow the study protocol orientations.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with obesity and diabetes
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of hypertension medication prescription | 12 months
  Reduction of hypertension medication prescription related to the baseline hypertension treatment at 12 months after surgery.

SECONDARY OUTCOMES:
Reduction of hypertension medication prescription | 1 month to 6 months
  Reduction of hypertension medication prescription compared to the baseline hypertension treatment at 1, 3 and 6 months.

OTHER OUTCOMES:
Change from baseline in systolic blood pressure | 1 to 12 months
Change from baseline in diastolic blood pressure | 1 to 12 months
Change from baseline in body weight | 1 to 12 months
Change from baseline in body mass index | 1 to 12 months
Change from baseline in waist circumference | 1 to 12 months
Change from baseline in body fat distribution | 1 to 12 months
Change from baseline in fasting plasma glucose | 1 to 12 months
Change from baseline in fasting plasma insulin | 1 to 12 months
Change from baseline in HbA1c | 3 to 12 months
Change from baseline in total cholesterol | 1 to 12 months
Change from baseline in LDL-cholesterol | 1 to 12 months
Change from baseline in HDL-cholesterol | 1 to 12 months
Change from baseline in triglycerides | 1 to 12 months
Change from baseline in artery vasodilative function | 1 to 12 months
  Endothelium-dependent nitroglycerin(NTG)-induced dilatation and flow-mediated dilatation (FMD) by non-invasive high-resolution ultrasound.
Change from baseline in serum amino acids level | 1 to 12 months
Change from baseline in sense of taste | 1 to 12 months
Change from baseline in hepatic enzymes | 1 to 12 months
Change from baseline in serum creatine | 1 to 12 months
Change from baseline in serum electrolyte | 1 to 12 months
Change from baseline in complete blood count | 1 to 12 months
Adverse events | 1 to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Military Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Sun F, Zhou X, Li Q, Li Y, Zhang H, Yan Z, He H, Zhao Z, Ke Z, Gao Y, Li F, Tong W, Zhu Z. Achieving blood pressure targets and antihypertensive effects through metabolic surgery in type 2 diabetes patients with hypertension. Diabetes Metab Res Rev. 2021 May;37(4):e3422. doi: 10.1002/dmrr.3422. Epub 2020 Nov 30. PMID 33197293